CLINICAL TRIAL: NCT07076862
Title: Multiparametric Total-Body [18F]F-AraG PET/CT Imaging in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: Multiparametric [18F]F-AraG Imaging in Post-Acute Sequelae of COVID-19 (PASC)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2339805; 1R01AI185685-01A1 (NIH)
Record Dates: First submitted 2025-07-10; First posted 2025-07-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: PASC Post Acute Sequelae of COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — 2,5-dichloro-4-bromophenol

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled into one of four parallel imaging subgroups based on disease status and study group assignment. No crossover will occur.
Masking Description: Thisis an open-label study. Neither participants nor investigators are blinded to imaging group assignment or visit schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A.1 - Control Group (90-min dynamic + 4-h static PET/CT) (Experimental): Control participants in this arm will undergo a 90-minute dynamic [¹⁸F]F-AraG total-body PET/CT scan, followed by a second 30-minute static PET/CT scan approximately 4 hours after tracer injection. Blood samples will be collected during the dynamic scan to support kinetic modeling.
  Interventions: Drug: A.1 - [¹⁸F]F-AraG PET/CT (90-min dynamic + 4-h static)
- A.2 - Control Group (60-min dynamic PET/CT only) (Experimental): Control participants in this arm will undergo a 60-minute dynamic [¹⁸F]F-AraG total-body PET/CT scan. No delayed imaging will be performed. Blood samples will be collected during the dynamic scan.
  Interventions: Drug: A.2 - [¹⁸F]F-AraG PET/CT (60-min dynamic only)
- B.1 - PASC Group (90-min dynamic + 4-h static PET/CT) (Experimental): PASC participants in this arm will undergo a 90-minute dynamic [¹⁸F]F-AraG total-body PET/CT scan, followed by a second 30-minute static scan approximately 4 hours post-injection. Blood samples are collected during the scan.
  Interventions: Drug: B.1 - [¹⁸F]F-AraG PET/CT (90-min dynamic + 4-h static)
- B.2 - PASC Group (60-min dynamic PET/CT only) (Experimental): PASC participants in this arm will undergo a 60-minute dynamic [¹⁸F]F-AraG PET/CT scan. No delayed imaging is performed. Blood samples are collected during imaging.
  Interventions: Drug: B.2 - [¹⁸F]F-AraG PET/CT (60-min dynamic only)

INTERVENTIONS:
Drug: A.1 - [¹⁸F]F-AraG PET/CT (90-min dynamic + 4-h static) — Participants receive an intravenous injection of 5 mCi (±20%) of [¹⁸F]F-AraG followed by a 90-minute total-body PET/CT scan and an additional 30-minute static scan at 4 hours post-injection. Blood samples (up to 42 mL total) are collected during dynamic imaging.
  Arms: A.1 - Control Group (90-min dynamic + 4-h static PET/CT)
Drug: A.2 - [¹⁸F]F-AraG PET/CT (60-min dynamic only) — Participants receive an intravenous injection of 5 mCi (±20%) of [¹⁸F]F-AraG followed by a 60-minute total-body PET/CT scan. Blood samples (up to 42 mL total) are collected during dynamic imaging.
  Arms: A.2 - Control Group (60-min dynamic PET/CT only)
Drug: B.1 - [¹⁸F]F-AraG PET/CT (90-min dynamic + 4-h static) — Participants receive an intravenous injection of 5 mCi (±20%) of [¹⁸F]F-AraG followed by a 90-minute total-body PET/CT scan and a second 30-minute scan at 4 hours. Blood samples (up to 42 mL total) are collected during dynamic imaging.
  Arms: B.1 - PASC Group (90-min dynamic + 4-h static PET/CT)
Drug: B.2 - [¹⁸F]F-AraG PET/CT (60-min dynamic only) — Participants receive 5 mCi (±20%) of [¹⁸F]F-AraG intravenously followed by a 60-minute total-body PET/CT scan. Blood samples (up to 42 mL total) are collected during dynamic imaging.
  Arms: B.2 - PASC Group (60-min dynamic PET/CT only)

SUMMARY:
This study uses total-body [¹⁸F]F-AraG PET/CT imaging to investigate immune activation and vascular changes in individuals with post-acute sequelae of SARS-CoV-2 infection (PASC), also known as Long COVID. Participants will undergo dynamic PET/CT imaging along with blood biomarker assessments and symptom evaluations. The study aims to characterize sites of immunological perturbation, correlate PET imaging findings with peripheral blood markers, and evaluate longitudinal changes in tissue-based immune activity in relation to symptom patterns over time. Data from this study will improve understanding of tissue-level immune dysregulation in PASC and support future clinical tools for assessing and managing this condition.

DETAILED DESCRIPTION:
Post-acute sequelae of SARS-CoV-2 infection (PASC) is associated with persistent immune dysregulation affecting multiple organ systems. This prospective, non-randomized, open-label research study will apply high-sensitivity total-body PET/CT imaging using the investigational radiotracer [¹⁸F]F-AraG to map immune activation across diverse tissues in PASC and COVID-19-recovered control participants. The tracer, [¹⁸F]F-AraG, selectively accumulates in activated T cells and allows kinetic modeling of immune cell activity in vivo.

A total of 51 participants will be enrolled, including 34 PASC participants and 17 controls. All participants will undergo baseline imaging, and a subset of 17 PASC participants will complete two additional follow-up scans at 4 and 8 months. Each imaging visit includes a dynamic PET/CT scan, peripheral blood draws for plasma proteomics and immunophenotyping, and symptom questionnaires collected through the UCSF LIINC cohort.

Findings will be used to identify tissue-specific immune signatures associated with symptom phenotypes and assess how these evolve over time. The results will help clarify the biological basis of PASC and support the development of future diagnostic or monitoring strategies. No direct health benefit is anticipated for participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Ability to understand the purposes and risks of the trial and willingness to sign an IRB-approved informed consent form.
3. Willingness and ability to comply with all protocol required procedures.
4. For participants of reproductive potential, defined as individuals who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months), or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy, willingness to use effective double barrier contraceptive methods (excluding withdrawal or timing methods) during the study and up to 1 day after the last administration of the radiotracer.
5. Previous diagnosis of SARS-CoV-2 infection as defined by a prior positive SARS-CoV-2 nucleic acid-based diagnostic test performed in a clinical laboratory on one or more nasopharyngeal or respiratory secretion samples or from an FDA-approved rapid antigen test at home. Documentation of the positive test will be requested but not required; if not available the participant will be asked to attest to the presence of a positive test.
6. Onset of COVID-19 symptoms (or if no symptoms, time of initial nucleic acid or antigen-based diagnostic test) at least 3 months prior to the baseline study visit.
7. Ability to travel to our research sites in San Francisco and Sacramento.
8. Laboratory evaluations obtained within 60 days prior to entry:

   1. Hemoglobin ≥ 8g/dL
   2. Platelet count ≥ 75,000 cells/mm3
   3. Absolute neutrophil count (ANC) > 1000 cells/mm3
   4. Aspartate aminotransferase (AST) < 3 × ULN units/L
   5. Alanine aminotransferase (ALT) < 3 × ULN units/L
   6. Calculated creatinine clearance (CrCl) ≥ 60mL/min as estimated by the Cockcroft-Gault equation:

   For men, (140 - age in years) × (body weight in kg) ÷ (serum creatinine in mg/dL × 72) = CrCl (mL/min)*

   *For women, multiply the result by 0.85 = CrCl (mL/min)
9. For PASC participants only: Reporting at least 2 unexplained symptoms, with at least 1 symptom in the fatigue domain and at least 1 symptom in either cardiopulmonary or neurocognitive domains, that last for at least 2 months and cannot be explained by an alternative diagnosis. Symptoms may be new onset after initial COVID-19 recovery or persist from the initial acute phase and may fluctuate or relapse over time. (According to World Health Organization definition of PASC http://www.WHO.int )
10. For control participants only: Individuals who have made full clinical recovery within 4-12 weeks of acute COVID-19 infection with no newly developed symptoms or changes in health after recovery.

Exclusion Criteria:

1. Serious comorbidities (nonmalignant disease or other conditions) that in the opinion of the investigator could compromise protocol objectives.
2. Any condition that alters the function of their immune system or any conditions caused by malfunction of their immune system and would interfere with imaging, including known underlying inflammatory or immune disorders, systemic malignancy, or other chronic viral infections (such as HIV, hepatitis B and hepatitis C).
3. Received vaccination of any type, including a SARS-CoV-2 vaccine, within 30 days of imaging
4. Pregnant or nursing individuals. A urine or HCG serum pregnancy test with a sensitivity of at least 25 mIU/mL will be performed at screening and on the day of PET/CT imaging at no charge to all participants of reproductive potential (see definition above).
5. Participants who have had prior allogeneic stem cell or solid organ transplant.
6. Previously diagnosed myelodysplasia syndrome or history of lymphoproliferative disease prior to study entry.
7. Active systemic autoimmune diseases not related to COVID-19.
8. Self-reported history of dysphoria or anxiety in closed spaces (i.e., uncontrolled claustrophobia).
9. Concurrent or prior enrollment in a separate research study involving a PET scan performed within the last 12 months for research purposes only.
10. Body weight is more than 240 kg (529 pounds)
11. Prisoners
12. Life expectancy < 24 months
13. Recent use of medication including guanosine or cysteine analogs.
14. Any other criteria which would make the participant unsuitable for enrollment to this study, as determined by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of [¹⁸F]F-AraG uptake kinetics in PASC and control participants | Baseline Imaging Visit
  To assess immune activation in convalescent COVID-19, dynamic PET/CT scans will be analyzed to generate time-activity curves (TACs) in multiple tissues. Kinetic modeling will be applied to extract uptake parameters including SUV, SUVR, Vt, Ki, and k3. These values will be reported and statistically compared between PASC and control participants.
Correlation between [¹⁸F]F-AraG uptake parameters and blood-based markers of immune dysregulation | Baseline imaging visit and baseline blood draw
  Spearman correlation tests and heat map clustering will be used to assess the association between PET-derived uptake measures and plasma biomarkers of inflammation and immune activation. Correlations will be examined in tissues showing significant uptake differences between study groups.
Longitudinal change in [¹⁸F]F-AraG uptake and correlation with PASC symptom scores | Baseline, 4-month, and 8-month follow-up visits (subset of PASC participants only)
  In a subset of participants, follow-up PET/CT imaging at 4 and 8 months will be used to assess within-subject change in kinetic uptake parameters. These changes will be compared to changes in symptom burden as measured by PHQ-15 symptom domain scores.

SECONDARY OUTCOMES:
Feasibility of blood flow kinetic modeling using early [¹⁸F]F-AraG dynamic PET data | Baseline imaging visit
  Early-phase TACs (< 5 min post-injection) will be fitted using the AATH model to estimate blood flow from the vascular phase of radiotracer distribution. Identifiability of kinetic parameters associated with vascular function will be evaluated. Mean values will be compared between study groups.
Correlation between vascular imaging parameters and blood biomarkers of vascular dysfunction | Baseline imaging visit and baseline blood draw
  Spearman correlations and heatmap analyses will be used to examine associations between PET-derived vascular parameters and plasma markers of vascular dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Negar Omidvari, PhD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UC Davis EXPLORER Molecular Imaging Center, Sacramento, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No